CLINICAL TRIAL: NCT05815615
Title: Study of the Side Effects of Plasmapheresis: a Multi-modal Approach
Brief Title: Plasmapheresis: a Multi-modal Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: RK2020
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Plasmapheresis; Haematology; Sport Performance; Body Composition; Inflammation; Immunology; Adverse Events
MeSH Terms: conditions — Inflammation | interventions — Plasmapheresis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): Simulated plasma donation, same procedure as for plasmapheresis but without drawing blood.
  Interventions: Device: Plasmapheresis
- Low-frequency (Experimental): Plasma donation 1x/month for 3 months
  Interventions: Device: Plasmapheresis
- High-frequency (Experimental): Plasma donation 3x/month for 3 months
  Interventions: Device: Plasmapheresis
- US scheme (Experimental): Plasma donation 2x/week for 3 months
  Interventions: Device: Plasmapheresis

INTERVENTIONS:
Device: Plasmapheresis — Plasma donation at different frequencies

SUMMARY:
Only very few studies have prospectively looked at the effect of repeated intensive plasma donation. In collaboration with the Rode Kruis Vlaanderen, we have recently found that repeated whole blood donation with a 3-month interval in between induced a drop in markers for iron status, which worsened with the number of donations. The repetition effect of the donations, whether whole blood or plasma, can be different from the effects measured after one single donation. It is therefore critical to test and document this repetitive effect to build trustable and valid guidelines concerning repetitive plasma donation.

ELIGIBILITY:
Inclusion criteria:

* male,
* age between 18-50 years
* BMI between 20-28 kg/m2
* aptitude to perform maximal physical efforts assessed by the physical activity readiness questionnaire (PAR-Q)

Exclusion criteria:

* The specific exclusion criteria of the Rode Kruis Vlaanderen for blood donation will not be systematically applied to the present study to increase the pool of recruitment.

  * In case the subjects do not comply with the criteria of the Rode Kruis Vlaanderen, their plasma donations will be thrown away.
  * In case the subjects comply, their plasma donations will be handled as usually.
* The criteria will be assessed before each plasma donation by a questionnaire as usually done in the Center of the Rode Kruis.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Blood markers | 3 months
  albumin in g/l
Blood markers | 3 months
  Immunoglobulins G, M and A in G/l
Sport performance | 3 months
  VO2max in mlO2/kg/min determined breath-by-breath on a cycloergometer
Sport performance | 3 months
  maximal force of the quadriceps in kg measured on a leg extension machine

SECONDARY OUTCOMES:
Body composition | 3 months
  fat mass in kg measured by DEXA
Body composition | 3 months
  lean mass in kg measured by DEXA
Blood pressure | 3 months
  systolic and diastolic blood pressure in mmHG

OTHER OUTCOMES:
Blood markers | 3 months
  red blood cells in 10^6/mm^3
Blood markers | 3 months
  haemoglobin in g/dl
Blood markers | 3 months
  haematocrit in %
Blood markers | 3 months
  iron in ug/dl
Blood markers | 3 months
  ferritin in ug/l
Blood markers | 3 months
  glycated haemoglobin in %
Blood markers | 3 months
  creatine kinase in U/l
Blood markers | 3 months
  total cholesterol in mg/dl
Blood markers | 3 months
  reticulocytes in %
Weight | 3 months
  in kg

CONTACTS AND LOCATIONS:
Locations (1):
- UCLouvain, Louvain-la-Neuve, Brabant Wallon, Belgium

IPD SHARING:
Plan to Share IPD: No